CLINICAL TRIAL: NCT02857894
Title: Identification of the Predisposing Genetic Factors of Idiopathic Polypoidal Vasculopathies in the ATM Gene (Ataxia Telangiectasia Mutated)
Brief Title: Genetic Factors of Idiopathic Polypoidal Vasculopathies in the ATM Gene (Ataxia Telangiectasia Mutated)
Acronym: ATM
Status: Terminated | Type: Observational
Why Stopped: Mutations found do not modify the ATM protein+ modifications of methodology would be necessary
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MMT_2015_4
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Choroidal Neovascularization
Keywords: Polypoidal choroidal vasculopathy
MeSH Terms: conditions — Choroidal Neovascularization; Polypoidal Choroidal Vasculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Polypoidal choriodal vasculopathy (PCV) is an ophthalmologic disease, characterized by vascular abnormalities of the walls of small choroidal vessels, reproducing the specific aspect of polyps (cluster aspect). PCV is one of the "boundary-forms" of age related macular degeneration.

These vasculopathies can be idiopathic. Following the radiotherapy treatments of active and occult-typed neovessels in Age-Related Macular Degeneration (ARMD), 10% of the patients would present typical polypoidal vasculopathic lesions. These polypoidal secondary lesions have been induced by radiotherapy treatment and may show an increased sensibility to radiation in these patients.

Such an increase of radiosensibility is noticed in ataxia telangiectasia syndrome, in relation to the ATM gene mutations. The secondary or idiopathic polypoidal vasculopathic lesions are to be brought closer to telangiectasias in Ataxia Telangiectasia. Considering the iatrogenic component of radiotherapy in the secondary forms of ataxia telangiectasia, it seems legitimate to search for predisposing variants to polypoidal vasculopathies in the ATM gene.

Considering the frequency of PCV worldwide, it seems important to identify the predisposing genetic factors of the ATM gene. These biomarkers to the pathology might enable us to offer prevention (reinforced protection against radiations, including light) and to develop therapeutics (recruitment of other kinases, ATM's partners, in the stability and cellular control of DNA).

ELIGIBILITY:
Inclusion Criteria:

* Adult caucasian patient
* Polypoidal choriodal vasculopathy
* Informed written consent

Exclusion Criteria:

* History of cephalic radiotherapy
* Absence of affiliation to social security or universal health coverage (CMU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with polypoidal choriodal vasculopathy
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
Variants in the ATM gene | Day 1
  Compared analysis of the variants frequency (heterozygote, homozygote variants versus the wild variant) in the ATM gene.

CONTACTS AND LOCATIONS:
Overall Officials: Martine MAUGET FAYSSE, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (1):
- Fondation Ophtalmologique A. de Rotchschild, Paris, France